CLINICAL TRIAL: NCT05089136
Title: Transcatheter Para-Valvular Leak Closure: An International Prospective Multicentre Registry
Acronym: FFPP1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: 16.622
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Valvular Heart Disease; Valve Disease, Heart
Keywords: cardiac valve; cardiac catheterization; paravalvular leak
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: transcatheter paravalvular leak closure — Transcatheter paravalvular leak closure (PVLc) was first described in 1992 and has since then emerged as an attractive alternative to repeat surgery. Many implantable devices that can be used for transcatheter PVLc have been marketed, although few are specifically designed for this purpose. It consist in implanting an occluder in the paravalvular leak to stop or reduce the regurgitant flow.

SUMMARY:
Prosthetic paravalvular leaks (PVL) leading to heart failure and/or haemolysis can be treated by interventional cardiology or open-heart surgery. Predictors of clinical success of transcatheter closure remains little known and should be identified to help choose between these two options.Patient selection criteria for the best option are needed. The investigators aimed to identify predictors of clinical success after transcatheter PVL closure. Consecutive patients referred to 24 European centres for transcatheter PVL closure in 2017-2019 were included in a prospective registry (Fermeture de Fuite ParaProthétique, FFPP) and followed over 2 years

DETAILED DESCRIPTION:
Prosthetic paravalvular leaks (PVL) are associated with congestive heart failure and haemolysis, for which the standard treatment is open-heart surgery with the attendant risks to the patient. Transcatheter closure has emerged as an alternative. Patient selection criteria for the best option are needed. The investigators aimed to identify predictors of clinical success after transcatheter PVL closure.

The investigators designed a prospective multicentre observational registry named Fermeture des Fuites Para-Prothétiques (FFPP, closure of PVLs). In Belgium, France, Poland, and Turkey, 24 centres each enrolled at least 1 patient, between 1 January, 2017 and 31 December, 2019. All centres included consecutive patients referred for PVL closure.

Patients were selected for transcatheter PVL closure as opposed to first-line surgical PVL closure if they were at high or prohibitive surgical risk or as an alternative option to surgery if transcatheter PVLc feasibility was high. Patients were selected by each heart-team of participating centre according to local practice.

The study was coordinated by the clinical research unit of the Marie Lannelongue Hospital (Le Plessis-Robinson, France) and was approved by an independent ethics committee (CCTIRS, 23 November 2016, n°16.622bis). It complied with the principles set forth in the Declaration of Helsinki. Informed and signed consent was obtained in all patients prior to the procedures.

Data collection An electronic case-report form (eCRF, Easy-crf.com) was completed for each patient. The medical history (notably regarding heart surgery), symptoms, physical findings, laboratory test results, and echocardiographic parameters were collected. The EUROSCORE II risk score (http://euroscore.org) was determined, since surgical valve replacement was among the treatment options. Creatinine clearance below 60 mL/min defined renal failure and below 30 mL/min severe renal failure. Heart failure was defined according to the European Society of Cardiology as the presence of symptoms (dyspnoea, orthopnoea, asthenia) with physical signs of heart failure (limb oedema, hepato-jugular reflux, crackles on pulmonary auscultation) linked to the valvular disease.20 Anaemia was defined as haemoglobin <13 g/dL in men and <12 g/dL in women and haemolytic anaemia as anaemia with lactic dehydrogenase elevation and/or schistocytes and/or low haptoglobin, in the absence of other causes of anaemia.

Definitions of technical and clinical success Both technical success and clinical success were defined according to the Paravalvular Leak Academic Research Consortium. Technical success was implantation of at least one device within the leak, with an at least 1-grade decrease in the echocardiographic leak-severity grade, no valve dysfunction, and no surgical conversion of the procedure. Clinical success was survival at one month without re-admission for heart failure, blood transfusion, or open-heart valvular surgery.

Adverse events The investigators recorded intra-procedural adverse events, in-hospital adverse events (during the index hospitalisation), and adverse events within the first month after the procedure. Adverse events occurring beyond the first month but during the index hospitalisation were classified as in-hospital adverse events.

Adverse event severity are graded using a five-level scale. Major adverse events were potentially life-threatening. Bleeding, haemolytic anaemia, acute kidney injury, vascular complications, and life-threatening events were defined according to the Paravalvular Leak Academic Research Consortium.

Prospective follow-up is performed over to year.The end of follow-up is expected on the 31th of december 2021

ELIGIBILITY:
Inclusion Criteria:

All centres included consecutive patients referred for PVLc. Patients were selected for transcatheter PVLc as opposed to first-line surgical PVLc if they were at high or prohibitive surgical risk or as an alternative option to surgery if transcatheter PVLc feasibility was high. Patients were selected by each heart-team of participating centre according to local practice.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An electronic case-report form (eCRF, Easy-crf.com) was completed for each patient. The medical history (notably regarding heart surgery), symptoms, physical findings, laboratory test results, and echocardiographic parameters were collected. The EUROSCORE II risk score (http://euroscore.org) was determined, since surgical valve replacement was among the treatment options. Creatinine clearance below 60 mL/min defined renal failure and below 30 mL/min severe renal failure. Heart failure was defined according to the European Society of Cardiology as the presence of symptoms (dyspnoea, orthopnoea, asthenia) with physical signs of heart failure (limb oedema, hepato-jugular reflux, crackles on pulmonary auscultation) linked to the valvular disease. Anaemia was defined as haemoglobin <13 g/dL in men and <12 g/dL in women and haemolytic anaemia as anaemia with lactic dehydrogenase elevation and/or schistocytes and/or low haptoglobin, in the absence of other causes of anaemia.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Death or secondary valve replacement | 2 years
  Rate of death or secondary valve replacement (transcatheter or surgical replacement)

SECONDARY OUTCOMES:
Hospitalization for heart failure | 2 years
  Number of hospitalization for heart failure after the procedure
Hemolysis | 2 years
  Number of hemolysis requiring blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Gerardin, Principal Investigator — Hopital Marie Lannelongue

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hascoet S, Smolka G, Blanchard D, Kloeckner M, Brochet E, Bouisset F, Leurent G, Thambo JB, Combes N, Dumonteil N, Bauer F, Nejjari M, Pilliere R, Dauphin C, Bonnet G, Ciobotaru V, Ketelers R, Gallet R, Hammoudi N, Mangin L, Bouvaist H, Spaulding C, Aminian A, Kilic T, Popovic B, Armero S, Champagnac D, Gerardin B. Predictors of Clinical Success After Transcatheter Paravalvular Leak Closure: An International Prospective Multicenter Registry. Circ Cardiovasc Interv. 2022 Oct;15(10):e012193. doi: 10.1161/CIRCINTERVENTIONS.122.012193. Epub 2022 Oct 18. PMID 36256693